CLINICAL TRIAL: NCT00111865
Title: Randomized Controlled Trial of Exercise in Lymphoma Patients
Brief Title: Healthy Exercise for Lymphoma Patients (HELP)
Acronym: HELP
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Lance Armstrong Foundation (Other)
Responsible Party: Kerry S. Courneya, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 04 Courneya
Record Dates: First submitted 2005-05-26; First posted 2005-05-27 (Estimated); Last update posted 2008-08-26 (Estimated); Status verified 2008-08

CONDITIONS: Lymphoma
Keywords: physical exercise; quality of life; lymphoma
MeSH Terms: conditions — Lymphoma; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise (Experimental): Aerobic Exercise Training
  Interventions: Behavioral: Aerobic Exercise Training
- Usual Care (No Intervention)

INTERVENTIONS:
Behavioral: Aerobic Exercise Training — The exercise group will perform supervised stationary cycle ergometer exercise 3 days/week for 12 weeks and be progressed from 15 to 45 minutes and 60% to 80% of their VO2 reserve over the course of the intervention.
  Arms: Exercise

SUMMARY:
Objectives: The primary objective of this trial is to determine the effect of aerobic exercise training (AET) on change in quality of life (QoL) in lymphoma survivors receiving and not receiving chemotherapy. Secondary objectives are to determine the effects of AET on changes in psychosocial outcomes, cardiopulmonary fitness, body composition, and treatment completion rates.

DETAILED DESCRIPTION:
Design and Setting: The study is a randomized controlled trial. It will be conducted at the University of Alberta and Cross Cancer Institute in Edmonton, Alberta, Canada.

Participants: Participants will be 120 lymphoma survivors diagnosed with either non-Hodgkin's lymphoma (NHL) or Hodgkin's disease (HD) and receiving or not receiving at least 8 weeks of chemotherapy at the Cross Cancer Institute in Edmonton, Alberta. Participants will be stratified by disease type (indolent NHL versus aggressive NHL versus HD) and planned chemotherapy protocol (no chemotherapy versus < 16 weeks versus > 16 weeks), and randomly assigned to either a 12 week exercise program or usual care.

Eligibility: Participants will be recruited from the Cross Cancer Institute. The eligibility criteria include medical, demographic, and logistic criterion, and are focused on internal validity as well as external validity. Eligibility criteria for the study are: (1) histologically confirmed lymphoma cancer, (2) 18 years of age or older, (3) not receiving chemotherapy or scheduled to receive at least 2 cycles (8 weeks) of chemotherapy, excluding high dose chemotherapy with stem cell transplant, (4) approval of the treating oncologist, (5) able to understand and provide written informed consent in English, (6) no uncontrolled hypertension, (7) no uncontrolled cardiac illness, (8) no active psychiatric condition, and (9) no contraindications to exercise as determined by a maximal fitness test conducted by a certified fitness consultant (CFC).

Recruitment: We have recruited 122 participants to the trial. The study is now closed to accrual.

Recruitment will take place at the treatment or follow-up consultation with the medical or radiation oncologist. Interested survivors will receive an information package from the oncologist and a follow-up telephone call from the project director who will explain the study further and answer any questions. All individuals who are interested in participating in the study will: (a) be asked to provide informed consent, (b) complete a self administered questionnaire, and (c) be scheduled for a maximal physical fitness test, a dual-x-ray absorptiometry (DEXA) scan, and a blood draw. The physical fitness test will determine final eligibility for the study.

Interventions: The exercise group will perform supervised stationary cycle ergometer exercise 3 days/week for 12 weeks and be progressed from 15 to 45 minutes and 60% to 80% of their VO2 reserve over the course of the intervention. The usual care group will be asked not to begin a structured exercise training program during the next 12 weeks and will receive the exercise for 4 weeks following the postintervention assessment.

End Points: The primary end point is change in the Trial Outcome Index of QoL between baseline and postintervention. QoL will be assessed by the Functional Assessment of Cancer Therapy-Anemia (FACT-An) scale (Trial Outcome Index: Physical Well-being, Functional Well-being and Anemia Subscales). Secondary end points are changes in psychosocial outcomes, cardiopulmonary fitness, body composition, and treatment completion rates. Cardiopulmonary fitness will be assessed by a graded exercise test using gas exchange analysis. Body composition will be assessed by body mass index and a DEXA scan. Treatment completion rates will be assessed as the number of chemotherapy cycles received divided by the number planned.

Sample Size: Sample size calculation is based on the primary end point. A clinically important difference (CID) in the TOI of the FACT-An is 6.0 points. Sixty participants in each group will allow us to detect a 10.0 point difference in between group changes with a power of .80 and a two-tailed a of .05 (standard deviation = 18.0 points).

ELIGIBILITY:
Inclusion Criteria:

* Non-hodgkin's lymphoma (including chronic lymphocytic leukemia) or Hodgkin's disease
* Approval of the treating oncologist
* Scheduled to receive no chemotherapy or chemotherapy for at least 8 weeks
* Able to understand and provide written informed consent in English
* 18+ years of age
* No uncontrolled hypertension, cardiac illness, psychiatric condition
* No contraindication to exercise as determined by a fitness test

Exclusion Criteria:

* Pregnant.
* Transplant candidate.
* Unwilling to accept randomization.
* Any medical condition that would be a contraindication to exercise. The clinicians will make this decision.
* Unwilling to travel to/participate in the exercise program as defined by the protocol.
* Planned/known absence of greater than 2 weeks during the intended study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2005-04; Primary Completion 2008-08 (Actual); Study Completion 2009-04 (Estimated)

PRIMARY OUTCOMES:
Change in QoL between baseline and postintervention. | 12 weeks

SECONDARY OUTCOMES:
Changes in cardiopulmonary fitness | 12 weeks
psychosocial outcomes | 12 weeks
body composition | 12 weeks
treatment completion rates | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kerry S Courneya, Ph.D., Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Courneya KS, Forbes CC, Trinh L, Sellar CM, Friedenreich CM, Reiman T. Patient satisfaction with participation in a randomized exercise trial: effects of randomization and a usual care posttrial exercise program. Clin Trials. 2013;10(6):959-66. doi: 10.1177/1740774513495985. Epub 2013 Aug 5. PMID 23918843
- [Derived] Courneya KS, Sellar CM, Trinh L, Forbes CC, Stevinson C, McNeely ML, Peddle-McIntyre CJ, Friedenreich CM, Reiman T. A randomized trial of aerobic exercise and sleep quality in lymphoma patients receiving chemotherapy or no treatments. Cancer Epidemiol Biomarkers Prev. 2012 Jun;21(6):887-94. doi: 10.1158/1055-9965.EPI-12-0075. Epub 2012 Apr 20. PMID 22523181
- [Derived] Courneya KS, Stevinson C, McNeely ML, Sellar CM, Friedenreich CM, Peddle-McIntyre CJ, Chua N, Reiman T. Effects of supervised exercise on motivational outcomes and longer-term behavior. Med Sci Sports Exerc. 2012 Mar;44(3):542-9. doi: 10.1249/MSS.0b013e3182301e06. PMID 21814149